CLINICAL TRIAL: NCT05810324
Title: The Performance of 18F-FAPI PET/CT in Patients With Various Types of Cancer
Brief Title: 18F-FAPI PET/CT in Patients With Various Types of Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jilin University (Other)
Responsible Party: Principal Investigator, Ji Bin, Doctor, Jilin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ChinaJapanUHJLU
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-FAPI (Experimental): Experimental: Experimental: 18F-FAPI Each subject receive a single intravenous injection of 18F-FAPI, and undergo PET/CT imaging within the specificed time.
  Interventions: Drug: 18F-FAPI

INTERVENTIONS:
Drug: 18F-FAPI — Each patient receive a single intravenous injection of 18F-FAPI, and undergo PET/CT scan within specified time.
  Other Names: FAPI

SUMMARY:
To evaluate the potential usefulness of 18F-FAPI positron emission tomography/computed tomography (PET/CT) for the diagnosis of primary and metastatic lesions in various types of cancer.

DETAILED DESCRIPTION:
Subjects with various types of cancer underwent 18F-FAPI PET/CT either for an initial assessment or for recurrence detection. Tumor uptake was quantified by the maximum standard uptake value (SUVmax). Using histopathology and follow-up as gold standard, the sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of 18F-FAPI PET/CT were calculated.

ELIGIBILITY:
Inclusion Criteria:

* patients with suspected or new diagnosed or previously treated malignant tumors (supporting evidence may include MRI, CT, tumor markers and pathology report);
* patients who had scheduled 18F-FAPI PET/CT scan; (iv)
* patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

* patients with non-malignant lesions;
* patients with pregnancy;
* the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | 1 year
  The sensitivity, specificity and accuracy of 18F-FAPI PET/CT were calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Ji, Principal Investigator — China-Japan Union Hospital, Jilin University
Locations (1):
- China-Japan Union Hospital, Changchun, Jilin, China